CLINICAL TRIAL: NCT03764072
Title: A Phase 2B Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel-design Study of the Efficacy and Safety of VX-150 for Acute Pain Following Bunionectomy
Brief Title: A Dose-ranging Study to Evaluate Efficacy and Safety of VX-150 in Subjects With Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX18-150-104
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Participants received placebo matched to VX-150 for 2 days.
  Interventions: Drug: Placebo
- VX-150 - Dose Level 1 (Experimental): Participants received VX-150 1500 milligrams (mg) as first dose, followed by VX-150 750 mg every 12 hours (q12h) for 2 days.
  Interventions: Drug: VX-150
- VX-150 - Dose Level 2 (Experimental): Participants received VX-150 1000 mg once daily (qd) for 2 days.
  Interventions: Drug: VX-150
- VX-150 - Dose Level 3 (Experimental): Participants received VX-150 500 mg q12h for 2 days.
  Interventions: Drug: VX-150
- VX-150 - Dose Level 4 (Experimental): Participants received VX-150 500 mg as first dose, followed by VX-150 250 mg q12h for 2 days.
  Interventions: Drug: VX-150
- VX-150 - Dose Level 5 (Experimental): Participants received VX-150 250 mg qd for 2 days.
  Interventions: Drug: VX-150

INTERVENTIONS:
Drug: VX-150 — Capsules for oral administration.
  Arms: VX-150 - Dose Level 1; VX-150 - Dose Level 2; VX-150 - Dose Level 3; VX-150 - Dose Level 4; VX-150 - Dose Level 5
Drug: Placebo — Capsules for oral administration.
  Arms: Placebo

SUMMARY:
This study will evaluate the dose-response relationship and safety of VX-150 in treating acute pain following bunionectomy.

ELIGIBILITY:
Key Inclusion Criteria:

Before surgery:

* Body mass index (BMI) of 18.0 to 38.0 kilogram per meter square (kg/m^2)
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair, without collateral procedures, under regional anesthesia (Mayo and popliteal sciatic block) not to include base wedge procedure

After surgery:

* Subject reported pain of greater than or equal to (>=) 4 on Numeric Pain Rating Scale (NPRS) and moderate or severe pain on the Verbal Categorical Rating Scale (VRS) within 9 hours after removal of the popliteal sciatic block on Day 1
* Subject is lucid and able to follow commands
* All analgesic guidelines were followed during and after the bunionectomy

Key Exclusion Criteria:

Before surgery:

* History in the past 10 years of malignancy, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
* History of abnormal laboratory results >=2.5*upper limit of normal (ULN)
* History of peripheral neuropathy
* A known or clinically suspected infection with human immunodeficiency virus or hepatitis B or C viruses
* Prior medical history of bunionectomy or other foot surgery on the index foot
* History of peptic ulcer disease, or intolerance or unwillingness to receive ibuprofen

After surgery:

* Subject had a type 3 deformity requiring a base wedge osteotomy or concomitant surgery

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Lotus Clinical Research, Pasadena, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Started | 46 | 42 | 44 | 45 | 46 | 27
Completed | 46 | 42 | 43 | 45 | 45 | 26
Not Completed | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal of consent (due to lack of efficacy) | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal of consent (for other reason) | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- VX-150 - Dose Level 1: Participants received VX-150 1500 mg as first dose, followed by VX-150 750 mg q12h for 2 days.
- VX-150 - Dose Level 2: Participants received VX-150 1000 mg qd for 2 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5 | Total
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (14.21) | 44.6 (13.03) | 44.7 (13.23) | 46.4 (12.18) | 47.2 (11.51) | 48.7 (12.92) | 46.2 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 40 | 39 | 40 | 21 | 217
  Male | 6 | 5 | 4 | 6 | 6 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 15 | 13 | 16 | 8 | 82
  Not Hispanic or Latino | 30 | 28 | 29 | 32 | 30 | 19 | 168
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 1 | 0 | 4
  Asian | 2 | 2 | 3 | 2 | 4 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 13 | 10 | 6 | 3 | 39
  White | 38 | 35 | 27 | 31 | 34 | 23 | 188
  More than one race | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pain Intensity at Baseline (at 0 hours) as Recorded on Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was recorded on 11-point ordinal NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain.
  units on a scale | 6.5 (1.8) | 7.0 (2.0) | 6.5 (1.8) | 6.6 (1.7) | 5.9 (1.3) | 6.9 (1.6) | 6.5 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of the Pain Intensity Difference as Recorded on Numeric Pain Rating Scale (NPRS) 0 to 24 Hours (SPID24) After First Dose
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPID24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 Hours After First Dose
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
units on a scale | 19.1 (49.7) | 37.3 (45.6) | 32.3 (51.2) | 30.5 (46.9) | 27.5 (37.8) | 28.3 (43.6)
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1 vs VX-150 - Dose Level 2 vs VX-150 - Dose Level 3 vs VX-150 - Dose Level 4 vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.2107, Multiple Comparison Procedure-Modelling — Dose response Model - Linear
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 1 vs VX-150 - Dose Level 2 vs VX-150 - Dose Level 3 vs VX-150 - Dose Level 4 vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.0766, Multiple Comparison Procedure-Modelling — Dose response Model - Emax
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 1 vs VX-150 - Dose Level 2 vs VX-150 - Dose Level 3 vs VX-150 - Dose Level 4 vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.0989, Multiple Comparison Procedure-Modelling — Dose response Model - Logistic
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 1 vs VX-150 - Dose Level 2 vs VX-150 - Dose Level 3 vs VX-150 - Dose Level 4 vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.0927, Multiple Comparison Procedure-Modelling — Dose-response Model - Sigmoid Emax

2. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference as Recorded on NPRS 0 to 48 Hours (SPID48) After First Dose
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0= no pain to 10= worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 Hours After First Dose
Population: FAS.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
units on a scale | 77.4 (105.2) | 112.5 (88.4) | 106.1 (109.6) | 101.5 (103.2) | 90.9 (81.9) | 100.0 (102.6)

3. Secondary Outcome: Proportion of Participants With at Least 30 Percent (%) Reduction in NPRS at 24 Hours After First Dose of VX-150 Versus Placebo
Description: Pain intensity was recorded on 11-point ordinal NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 30% reduction from baseline in NPRS at 24 hours after the first dose of VX-150 or placebo were reported.
Time Frame: From Baseline at 24 Hours After First Dose
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
percentage of participants | 50.0 | 59.5 | 56.8 | 55.6 | 63.0 | 51.9
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1; Test type: Superiority; p = 0.3162, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 2; Test type: Superiority; p = 0.4613, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 3; Test type: Superiority; p = 0.4095, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 4; Test type: Superiority; p = 0.1570, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.9843, Cochran-Mantel-Haenszel

4. Secondary Outcome: Proportion of Participants With at Least 50% Reduction in NPRS at 24 Hours After the First Dose of VX-150 Versus Placebo
Description: Pain intensity was recorded on 11-point ordinal NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain. The percentage of participants with at least 50% reduction from baseline in NPRS at 24 hours after the first dose of VX-150 or placebo were reported.
Time Frame: From Baseline at 24 Hours After First Dose
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
percentage of participants | 41.3 | 38.1 | 45.5 | 44.4 | 45.7 | 40.7
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1; Test type: Superiority; p = 0.8714, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 2; Test type: Superiority; p = 0.5815, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 3; Test type: Superiority; p = 0.4308, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 4; Test type: Superiority; p = 0.4434, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.8550, Cochran-Mantel-Haenszel

5. Secondary Outcome: Proportion of Participants With at Least 70% Reduction in NPRS at 24 Hours After the First Dose of VX-150 Versus Placebo
Description: Pain intensity was recorded on 11-point ordinal NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain. The percentage of participants with at least 70% reduction from baseline in NPRS at 24 hours after the first dose of VX-150 or placebo were reported.
Time Frame: From Baseline at 24 Hours After First Dose
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
percentage of participants | 21.7 | 21.4 | 34.1 | 22.2 | 30.4 | 18.5
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1; Test type: Superiority; p = 0.6870, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 2; Test type: Superiority; p = 0.1515, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 3; Test type: Superiority; p = 0.6030, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 4; Test type: Superiority; p = 0.1361, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.5640, Cochran-Mantel-Haenszel

6. Secondary Outcome: Time to Onset of Confirmed Perceptible Pain Relief After First Dose of VX-150 Versus Placebo
Description: Time to onset of confirmed perceptible pain relief (time to onset of perceptible pain relief [any pain relief at all after the first dose] for participants who had meaningful pain relief [relief that is meaningful to participants after the first dose] reported based on the stopwatch assessment.
Time Frame: Up to 6 hours After the First Dose
Population: FAS.
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
minutes | 20.4 [6 to 67] | 29.6 [6 to 115] | 23.8 [11 to 92] | 20.2 [7 to 103] | 35.6 [2 to 112] | 25.2 [17 to 102]
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1; Test type: Superiority; p = 0.5405, Regression, Cox; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.60 to 2.67]
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 2; Test type: Superiority; p = 0.9011, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.49 to 2.27]
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 3; Test type: Superiority; p = 0.9127, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.48 to 2.26]
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 4; Test type: Superiority; p = 0.5619, Regression, Cox; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.60 to 2.56]
Statistical Analysis 5: Comparison: Placebo vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.7090, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.50 to 2.79]

7. Secondary Outcome: Time to Onset of Meaningful Pain Relief After the First Dose of VX-150 Versus Placebo
Description: Time to onset of meaningful pain relief (relief that is meaningful to participants after the first dose) reported based on the stopwatch assessment.
Time Frame: Up to 6 Hours After the First Dose
Population: FAS.
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
minutes | 55.4 [19 to 102] | 58.7 [16 to 175] | 68.6 [15 to 255] | 49.9 [20 to 355] | 61.5 [10 to 294] | 64.5 [30 to 162]
Statistical Analysis 1: Comparison: Placebo vs VX-150 - Dose Level 1; Test type: Superiority; p = 0.5141, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.61 to 2.72]
Statistical Analysis 2: Comparison: Placebo vs VX-150 - Dose Level 2; Test type: Superiority; p = 0.9614, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.45 to 2.12]
Statistical Analysis 3: Comparison: Placebo vs VX-150 - Dose Level 3; Test type: Superiority; p = 0.9756, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.46 to 2.14]
Statistical Analysis 4: Comparison: Placebo vs VX-150 - Dose Level 4; Test type: Superiority; p = 0.5582, Regression, Cox; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.60 to 2.57]
Statistical Analysis 5: Comparison: Placebo vs VX-150 - Dose Level 5; Test type: Superiority; p = 0.7543, Regression, Cox; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.49 to 2.71]

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of VRT- 1207355 (Active Moiety) and VRT- 1268114 (Metabolite M5)
Time Frame: Day 1 and Day 2
Population: Pharmacokinetic (PK) set included all randomized participants who received at least 1 dose of study drug. Here, "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 42 | 44 | 45 | 46 | 27
micrograms per milliliter (mcg/mL)
  VRT- 1207355: Day 1: number analyzed (Participants) | 41 | 40 | 43 | 43 | 24
  VRT- 1207355: Day 1 | 4.97 (1.67) | 3.27 (1.35) | 1.71 (0.536) | 1.89 (0.641) | 0.794 (0.241)
  VRT- 1207355: Day 2: number analyzed (Participants) | 39 | 39 | 42 | 44 | 23
  VRT- 1207355: Day 2 | 4.93 (1.38) | 4.17 (1.53) | 3.00 (0.979) | 1.95 (0.708) | 0.974 (0.305)
  VRT- 1268114: Day 1: number analyzed (Participants) | 41 | 39 | 43 | 43 | 24
  VRT- 1268114: Day 1 | 1.79 (0.637) | 1.31 (0.602) | 0.699 (0.261) | 0.719 (0.341) | 0.295 (0.128)
  VRT- 1268114: Day 2: number analyzed (Participants) | 39 | 39 | 42 | 44 | 23
  VRT- 1268114: Day 2 | 2.68 (0.944) | 1.87 (0.779) | 1.65 (0.544) | 1.11 (0.437) | 0.408 (0.153)

9. Secondary Outcome: Area Under the Concentration Versus Time Curve From 0 to 12 Hours (AUC0-12h) of VRT- 1207355 and VRT- 1268114
Time Frame: Day 1 and Day 2
Population: PK set. Here, "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 42 | 44 | 45 | 46 | 27
microgram*hour per milliliter (mcg*h/mL)
  VRT- 1207355: Day 1: number analyzed (Participants) | 40 | 40 | 42 | 43 | 24
  VRT- 1207355: Day 1 | 39.7 (13.4) | 25.7 (11.0) | 13.6 (4.60) | 14.6 (4.73) | 5.99 (1.68)
  VRT- 1207355: Day 2: number analyzed (Participants) | 39 | 39 | 42 | 44 | 23
  VRT- 1207355: Day 2 | 46.1 (14.0) | 36.1 (12.8) | 27.1 (8.40) | 17.7 (6.01) | 8.24 (2.80)
  VRT- 1268114: Day 1: number analyzed (Participants) | 40 | 39 | 42 | 43 | 24
  VRT- 1268114: Day 1 | 13.7 (4.40) | 10.2 (4.84) | 5.55 (2.04) | 5.48 (2.58) | 2.27 (1.01)
  VRT- 1268114: Day 2: number analyzed (Participants) | 39 | 39 | 42 | 44 | 23
  VRT- 1268114: Day 2 | 26.8 (9.60) | 17.6 (7.33) | 16.2 (4.72) | 10.8 (4.19) | 3.84 (1.39)

10. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 10
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
Number analyzed (Participants) | 46 | 42 | 44 | 45 | 46 | 27
participants
  Participants With AEs | 15 | 16 | 19 | 18 | 19 | 12
  Participants With SAEs | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 10
Arm/Group | Placebo | VX-150 - Dose Level 1 | VX-150 - Dose Level 2 | VX-150 - Dose Level 3 | VX-150 - Dose Level 4 | VX-150 - Dose Level 5
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/42 | 0/44 | 0/45 | 0/46 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/42 | 0/44 | 0/45 | 0/46 | 1/27
Other Adverse Events (participants affected / at risk) | 7/46 | 9/42 | 13/44 | 12/45 | 12/46 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | VX-150 - Dose Level 1 (N=42) | VX-150 - Dose Level 2 (N=44) | VX-150 - Dose Level 3 (N=45) | VX-150 - Dose Level 4 (N=46) | VX-150 - Dose Level 5 (N=27)
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | VX-150 - Dose Level 1 (N=42) | VX-150 - Dose Level 2 (N=44) | VX-150 - Dose Level 3 (N=45) | VX-150 - Dose Level 4 (N=46) | VX-150 - Dose Level 5 (N=27)
Headache (Nervous system disorders) | 5 | 7 | 9 | 8 | 8 | 2
Nausea (Gastrointestinal disorders) | 3 | 4 | 5 | 5 | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT03764072/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT03764072/SAP_001.pdf